CLINICAL TRIAL: NCT03620279
Title: Magic Camp for Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, principal investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001044
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: motor training for cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magic camp intervention (Experimental): These children are diagnosed with cerebral palsy and we will provide motor control training.
  Interventions: Behavioral: Magic camp intervention

INTERVENTIONS:
Behavioral: Magic camp intervention — Hand-arm bimanual motor skills training

SUMMARY:
The proposed study will test the feasibility and effectiveness of a "Magic Camp" in children with spastic hemiplegic cerebral palsy (CP). A single group pretest-posttest design (n=10) will be used to investigate the immediate (2 weeks) and longer-term effect (3 months) of a "Magic Camp" on improving upper limb motor function and health-related quality of life (HRQoL) in children with hemiplegic CP.

DETAILED DESCRIPTION:
This project will employ a single group pretest-posttest design to investigate the impact of a "Magic Camp" on the improvement in upper limb motor function, health-related quality of life, and emotional stress among children with spastic hemiplegic CP. After the baseline evaluation, eligible participants will complete one-on-one "magic trick" training 3-hours per day for 2 consecutive weeks. The primary outcome measures will be unimanual function as measured by the Jebsen Taylor Test of Hand Function, bimanual coordination as measured by kinematic parameters using motion analysis, and spontaneous use of the more affected limb in real-life activities that demand the use of both hands as measured by the Children's Hand Experience Questionnaire. Secondary outcome measures will include HRQoL as measured by the Cerebral Palsy Quality of Life Questionnaire, in-depth dyad qualitative interviews of the caregivers and children, and emotional stress as measured by the fingernail cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* spasticity with Modified Ashworth Scale grades between 1 and 3;
* ability to lift the more affected arm 15 cm above a table surface;
* impairment of hand function at levels I to III of the Manual Activity Classification System
* ability to grasp and release light objects with the more affected hand
* largely nonuse of the more affected hand in daily activities as determined by the Pediatric Motor Activity Log
* are interested in learning magic tricks
* have the cognitive and social ability to participate in a camp setting;
* ability to follow directions in English; and
* ability to remember simple sequences of actions to perform magic tricks.

Exclusion Criteria:

* severe muscle spasticity or fixed contracture in the more affected limb that limits functional arm and hand use
* dystonia
* severe visual or auditory disorders that prevent learning and carrying out the magic tricks
* serious or recurring medical complications
* participation in intensive upper limb intervention and/or musculoskeletal and tone management treatments, dorsal rhizotomy, or surgery on the upper limb in the previous 6 months or anticipated within subsequent 6 months
* start muscle relaxant within the last 3 months; or
* plan to move to another state within the next 6 months.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Unimanual skill as measured by the Jebsen Taylor Test of Hand Function | baseline
  Jebsen Taylor Test of Hand Function (JTTHF) is a standardized timed test administered by occupational therapy (OT) students to assess the efficiency of unimanual grasp and release of items with six tasks. Higher scores (i.e., longer duration the participant takes to complete the task) represent poorer unimanual skills
Bimanual coordination as measured by 3-D kinematic motion analysis | baseline
  Participants will be asked to perform the task with their preferred hand choice at a self-selected pace following by an auditory go-signal. Each trial ends when the button is pressed. Five trials will be collected after 2 practice trials, and outcome measures will be averaged over the 5 trials. Longer time duration it takes for the participant to complete the task represents poorer bimanual coordination.
Extent of the more affected hand use in daily bimanual activities as measured by the Children's Hand Experience Questionnaire (CHEQ) | Baseline
  CHEQ is a 29-item (parent and child report) questionnaire that evaluates the experience of children in using the more affected hand in activities where usually two hands are required. Percentage use of the more affected hand will be expressed as percentage of independent activities performed bimanually in which the more affected hand is used to stabilize or grip items. Higher percentage (ranging from 0% to 100%) represents higher extent of using the more affected hand.
Health-related quality of life as measured by the Cerebral Palsy Quality of Life (CPQOL) Questionnaire | Baseline
  CPQOL evaluates the well-being of children with CP across several broad domains such as social well-being and acceptance, and emotional well-being. Items are rated on a 9-point scale, and recoded and transformed into scaled scores (transformed to a scale of 1-100) for each domain. An average of the scale scores from all domains (family & friends, school, communication, health, special equipment, pain and bother, and access to services) is conducted. Higher scores represent better health-related quality of life.
Emotional stress as measured by the amount of cortisol in participants' and their caregivers' fingernails. | Baseline
  Fingernail samples from every digit will be collected by clipping directly into a Ziploc® bag to avoid losing any parts of the sample. Nail samples will be sent to the Bio-Analytical Redox Biology (BARB) Core Laboratory, University of Alabama at Birmingham (UAB) for analysis.

SECONDARY OUTCOMES:
Unimanual skill as measured by the Jebsen Taylor Test of Hand Function | from baseline to two weeks
  Jebsen Taylor Test of Hand Function (JTTHF) is a standardized timed test administered by OT students to assess the efficiency of unimanual grasp and release of items with six tasks. Higher scores (i.e., longer duration the participant takes to complete the task) represent poorer unimanual skills.
Bimanual coordination as measured by 3-D kinematic motion analysis | from baseline to two weeks
  Participants will be asked to perform the task with their preferred hand choice at a self-selected pace following by an auditory go-signal. Each trial ends when the button is pressed. Five trials will be collected after 2 practice trials, and outcome measures will be averaged over the 5 trials.Longer time duration it takes for the participant to complete the task represents poorer bimanual coordination.
Extent of the more affected hand use in daily bimanual activities as measured by the Children's Hand Experience Questionnaire (CHEQ) | from baseline to two weeks
  CHEQ is a 29-item (parent and child report) questionnaire that evaluates the experience of children in using the more affected hand in activities where usually two hands are required. Percentage use of the more affected hand will be expressed as percentage of independent activities performed bimanually in which the more affected hand is used to stabilize or grip items. Higher percentage (ranging from 0% to 100%) represents higher extent of using the more affected hand.
Health-related quality of life as measured by the Cerebral Palsy Quality of Life (CPQOL) Questionnaire | from baseline to two weeks
  CPQOL evaluates the well-being of children with CP across several broad domains such as social well-being and acceptance, and emotional well-being. Items are rated on a 9-point scale, and recoded and transformed into scaled scores for each domain. An average of the scale scores from all domains (family & friends, school, communication, health, special equipment, pain and bother, and access to services) is conducted. Higher scores represent better health-related quality of life.
Unimanual skill as measured by the Jebsen Taylor Test of Hand Function | from two weeks to three months
  Jebsen Taylor Test of Hand Function (JTTHF) is a standardized timed test administered by OT students to assess the efficiency of unimanual grasp and release of items with six tasks. Higher scores (i.e., longer duration the participant takes to complete the task) represent poorer unimanual skills.
Bimanual coordination as measured by 3-D kinematic motion analysis | from two weeks to three months
  Participants will be asked to perform the task with their preferred hand choice at a self-selected pace following by an auditory go-signal. Each trial ends when the button is pressed. Five trials will be collected after 2 practice trials, and outcome measures will be averaged over the 5 trials. Longer time duration it takes for the participant to complete the task represents poorer bimanual coordination.
Extent of the more affected hand use in daily bimanual activities as measured by the Children's Hand Experience Questionnaire (CHEQ) | from two weeks to three months
  CHEQ is a 29-item (parent and child report) questionnaire that evaluates the experience of children in using the more affected hand in activities where usually two hands are required. Percentage use of the more affected hand will be expressed as percentage of independent activities performed bimanually in which the more affected hand is used to stabilize or grip items. Higher percentage (ranging from 0% to 100%) represents higher extent of using the more affected hand.
Health-related quality of life as measured by the Cerebral Palsy Quality of Life (CPQOL) Questionnaire | from two weeks to three months
  CPQOL evaluates the well-being of children with CP across several broad domains such as social well-being and acceptance, and emotional well-being. Items are rated on a 9-point scale, and recoded and transformed into scaled scores for each domain. An average of the scale scores from all domains (family & friends, school, communication, health, special equipment, pain and bother, and access to services) is conducted. Higher scores represent better health-related quality of life.
Emotional stress as measured by the amount of cortisol in participants' and their caregivers' fingernails. | from baseline to three months
  Fingernail samples from every digit will be collected by clipping directly into a Ziploc® bag to avoid losing any parts of the sample. Nail samples will be sent to the BARB Core Laboratory, UAB for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hon K Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No